CLINICAL TRIAL: NCT07329959
Title: Safety and Efficacy of Immunosuppressive CAR-DC Targeting FAP in the Treatment of End-stage Idiopathic Pulmonary Fibrosis
Brief Title: CAR-DC for End-Stage IPF
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1161
Record Dates: First submitted 2025-12-07; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis(IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-DC Treatment (Experimental): Subjects aged 18-75 with end-stage IPF meeting eligibility criteria will be enrolled. The study comprises:
  1. Screening: Post-Informed Consent Form (ICF) signing, subjects are screened for eligibility. Only qualified subjects proceed.
  2. Leukapheresis: Hospitalized subjects undergo ~100 ml blood collection via apheresis. Valid infectious disease testing is required.
  3. Treatment: Hospitalized subjects receive a single infusion of autologous FAP-targeted iCDC cells. Pre-infusion criteria must be met (e.g., no significant infection, creatinine <2×ULN).
  4. Post-Treatment Evaluation: Outpatient visits at Months 1, 3, and 6 post-infusion (Day 0). Assessments include pulmonary function tests, chest CT, 6-minute walk test, physical exams, vital signs, lab tests, and peripheral blood monitoring for iCDC cells.
  5. Long-Term Follow-Up: For overall survival and long-term safety monitoring.
  Interventions: Procedure: Leukapheresis; Biological: CAR-DC

INTERVENTIONS:
Procedure: Leukapheresis — Subjects will be hospitalized in the Lung Transplant Ward to undergo leukapheresis, followed by an observation period. Eligible subjects, after signing the specific leukapheresis consent form, will undergo apheresis for the collection of approximately 100 ml of blood using a blood cell separator for the preparation of CAR-DC reagents.
Biological: CAR-DC — Subjects will be hospitalized to receive autologous FAP-targeted immunosuppressive CAR-DC cell therapy, followed by an observation period. Based on our team's preclinical studies, the starting dose was determined to be 4×10⁵ cells/kg. This trial will employ a standard "3+3" dose-escalation design: Dose Level -1 at 1×10⁵ cells/kg, Dose Level 1 (starting dose) at 4×10⁵ cells/kg, and Dose Level 2 at 8×10⁵ cells/kg.
  The 3+3 dose escalation begins with the Dose Level 1 administered to a cohort of three subjects. If no dose-limiting toxicities (DLTs) are observed, the dose is escalated for the next cohort. If one DLT occurs, the cohort is expanded to six subjects at the same dose; escalation proceeds only if no further DLTs are seen in the expanded cohort. If two or more DLTs occur at any point within a cohort, dose escalation stops, and the maximum tolerated dose (MTD) is defined as the highest dose level with an observed DLT rate of less than 2 out of 6 subjects.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic, progressive, fatal interstitial lung disease characterized by irreversible scarring, leading to respiratory failure. With limited treatment options and a poor prognosis, new therapies are urgently needed. This study investigates a novel cell therapy targeting pathological fibroblasts, a key driver of fibrosis.

Single-cell analyses identify CTHRC1+FAP+ fibroblasts as a collagen-producing subpopulation crucial in IPF progression. Chimeric antigen receptor (CAR) technology enables precise targeting of these cells. While CAR-Treg therapy has shown promise in preclinical models, its clinical translation requires careful safety evaluation regarding infection risk, potential tumor promotion, and immune reconstitution.

This trial employs an innovative approach using engineered dendritic cells (DCs). CAR technology is applied to generate immunosuppressive CAR-DCs (iCAR-DCs) designed to target FAP, localize to fibrotic lung areas, and attenuate fibrosis without eliciting a detrimental immune response. Preliminary mouse studies demonstrated that iCAR-DC administration following lung injury significantly reduced fibrosis without apparent organ toxicity and improved survival.

This single-arm trial aims to evaluate the efficacy and safety of this immunosuppressive CAR-DC therapy in patients with end-stage IPF. Key assessments will include changes in lung function, fibrosis extent on imaging, and comprehensive monitoring of potential adverse effects, particularly infections, tumor markers, and immune parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years, inclusive, with a diagnosis of idiopathic pulmonary fibrosis (IPF).

2. Ability to verbally confirm understanding of the risks, benefits, and alternative treatments associated with immunosuppressive CAR-DC therapy. Provision of written informed consent by the patient or their legally authorized representative prior to participation.

3. Evidence of disease progression (worsening pulmonary fibrosis and declining lung function) despite treatment with standard therapies such as pirfenidone, nintedanib, or other appropriate regimens.

4. Meets at least one criterion indicating eligibility for lung transplantation due to interstitial lung disease, while not consenting to a transplant. The criteria include:

1. A decline in forced vital capacity (FVC) ≥10% over a 6-month follow-up period.
2. A decline in diffusing capacity of the lungs for carbon monoxide (DLCO) ≥10% of predicted value over 6 months.
3. Six-minute walk test results showing oxygen saturation <88%, a distance walked <250 meters, or a decline of >50 meters in distance over 6 months.
4. Presence of pulmonary hypertension (PH) confirmed by right heart catheterization or transthoracic echocardiography.
5. Hospitalization due to respiratory functional decline, pneumothorax, or acute exacerbation.

5. No prior cellular immunotherapy within the last 3 months. 6. Hematological parameters meeting the following thresholds: hematocrit >30%, lymphocyte count >0.5 × 10⁹/L, and platelet count >60 × 10⁹/L.

Exclusion Criteria:

1. History of acute exacerbation of IPF within 4 weeks prior to screening or during the screening period.
2. Presence of interstitial lung disease (ILD) other than IPF, including but not limited to: other forms of idiopathic interstitial pneumonia; ILD associated with fibrogenic agents, environmental exposures, or drug toxicity; other occupational lung diseases; granulomatous lung diseases; pulmonary vascular diseases; or ILD related to systemic diseases (e.g., vasculitis, infections such as tuberculosis, connective tissue diseases). Cases with uncertain diagnosis require serological testing and/or multidisciplinary team review for confirmation.
3. Presence of significant active infection.
4. History of malignancy, except for malignancies treated with curative intent and with no recurrence for ≥5 years, resected basal cell or squamous cell skin carcinoma, carcinoma in situ of the cervix, or resected colonic polyps.
5. Significant history of infectious diseases.
6. Presence of psychiatric illness or other conditions that would compromise the patient's ability to cooperate with study requirements, comply with treatment, or undergo monitoring.
7. Known hypersensitivity to any component of the immunosuppressive CAR-DC cell product.
8. History of severe renal failure requiring renal dialysis, or serum creatinine level >2.5 mg/dL.
9. Any contraindication to the investigational product or study procedures.
10. Pregnancy or lactation.
11. History of pulmonary embolism (PE), deep vein thrombosis (DVT), or recurrent thromboembolic events.
12. Uncorrected thrombocytopenia (platelet count <50,000/μL) or systemic coagulopathy (INR >2.5 or aPTT >2.5 times the control value in the absence of anticoagulant therapy), or active bleeding with uncorrectable coagulopathy.
13. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels >5.0 times the upper limit of normal (ULN), or total bilirubin >3 mg/dL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
The safety and efficacy of targeted FAP immunosuppressive CAR-DC in the treatment of end-stage idiopathic pulmonary fibrosis | Within six months after CAR-DC therapy
  The incidence of dose-limiting toxicity (DLT) and treatment-related adverse events (TEAE) within 14 days was evaluated in the targeted FAP immunosuppressive CAR-DC therapy for end-stage idiopathic pulmonary fibrosis.

SECONDARY OUTCOMES:
The difference in forced vital capacity compared to the baseline before treatment | The three time points following CAR-DC cell therapy: Month 1, Month 3, and Month 6.
The difference in pulmonary carbon monoxide diffusion capacity compared to the baseline before treatment | The three time points following CAR-DC cell therapy: Month 1, Month 3, and Month 6.
The difference between the ratio of forced expiratory volume in the first second and forced vital capacity compared to the baseline before treatment | The three time points following CAR-DC cell therapy: Month 1, Month 3, and Month 6.
The difference between the 6-minute walk test result and the baseline value before treatment | The three time points following CAR-DC cell therapy: Month 1, Month 3, and Month 6.
The difference in the rate of change of pulmonary fibrosis area compared to the baseline before treatment as measured by quantitative CT | The three time points following CAR-DC cell therapy: Month 1, Month 3, and Month 6.
The total score of the St. George's Respiratory Questionnaire compared to the baseline before treatment | The three time points following CAR-DC cell therapy: Month 1, Month 3, and Month 6.
The total score of the MRC Questionnaire compared to the baseline before treatment. | The three time points following CAR-DC cell therapy: Month 1, Month 3, and Month 6.
The times of the acute exacerbation of IPF | Within six months after CAR-DC therapy
Number of participants with a set of laboratory tests | The seven time points following CAR-DC cell therapy: Day 0, Day 3, Day 7, Day 14, Month 1, Month 3, and Month 6.
  Blood biochemistry, commonly referred to as clinical chemistry or serum chemistry, is a foundational set of laboratory tests that quantitatively measures key chemical substances within the blood. It provides a vital snapshot of the body's metabolic state and the functional health of major organ systems.
Complete Blood Count | The seven time points following CAR-DC cell therapy: Day 0, Day 3, Day 7, Day 14, Month 1, Month 3, and Month 6.
  A complete blood count (CBC), often referred to as hematology in a clinical lab context, is one of the most fundamental and frequently ordered blood tests. It provides a quantitative and qualitative analysis of the cellular components of the blood.
Lymphocyte subpopulation detection | The seven time points following CAR-DC cell therapy: Day 0, Day 3, Day 7, Day 14, Month 1, Month 3, and Month 6.
  The proportion of each subgroup of lymphocytes in the subjects' blood was detected by flow cytometry.
Cytokine levels | The seven time points following CAR-DC cell therapy: Day 0, Day 3, Day 7, Day 14, Month 1, Month 3, and Month 6.
  The levels of cytokines such as IL2, IL4 and IL6 in the peripheral blood serum of the subjects were detected by ELISA method.
C-reactive protein | The seven time points following CAR-DC cell therapy: Day 0, Day 3, Day 7, Day 14, Month 1, Month 3, and Month 6.
  C-reactive protein (CRP) is a key acute-phase reactant and a non-specific but highly sensitive biomarker of systemic inflammation. Primarily produced by the liver in response to pro-inflammatory cytokines, its level in the blood rises rapidly in the presence of acute inflammation, infection, or tissue injury.
CAR gene copy number | The seven time points following CAR-DC cell therapy: Day 0, Day 3, Day 7, Day 14, Month 1, Month 3, and Month 6.
  CAR gene copy number refers to the average number of CAR transgene copies integrated into the genome of a patient's engineered T cells. Monitoring this parameter is critical in CAR-T cell therapy for both safety and efficacy reasons. This indicator will be detected by qPCR.

IPD SHARING:
Plan to Share IPD: No